CLINICAL TRIAL: NCT00961896
Title: A Double-blind, Randomized, Vehicle-controlled Proof of Concept (PoC) Study to Evaluate the Safety, Local Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Topical Administrations of LDE225 (a Specific Smoothened Inhibitor) on Skin Basal Cell Carcinomas in Gorlin Syndrome Patients Followed by an Open Label, Randomized Expansion Group to Test Two Different Strengths of an Improved LDE225 Formulation for Extended Treatment Durations
Brief Title: A Trial to Evaluate the Safety, Local Tolerability, Pharmacokinetics and Pharmacodynamics of LDE225 on Skin Basal Cell Carcinomas in Gorlin Syndrome Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLDE225B2203; EudraCT 2008 005506-40
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Results first posted 2015-09-21 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Treatment for Basal Cell Carcinomas (BCCs) in Gorlin Syndrome Patients
Keywords: Basal Cell Carcinoma; Gorlin Syndrome,; Gorlin-Goltz Syndrome,; Basal Cell Nevus Syndrome,; Nevoid Basal Cell Carcinoma Syndrome,; Basal Cell Carcinoma Nevus Syndrome
MeSH Terms: conditions — Carcinoma, Basal Cell; Basal Cell Nevus Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- LDE225 (applied in parallel with vehicle) [Part I] (Active Comparator): Participants were exposed to both topically applied 0.75% LDE225 cream and LDE225 vehicle cream twice daily for 28 days where each treatment was randomized to two different test areas on each participant.
  Interventions: Drug: LDE225 0.75%
- Vehicle cream (applied in parallel with LDE225 [Part I] (Placebo Comparator): Participants were exposed to both topically applied 0.75% LDE225 cream and LDE225 vehicle cream twice daily for 28 days where each treatment was randomized to two different test areas on each participant.
  Interventions: Drug: Vehicle
- LDE225 0.25% [Part II] (Active Comparator): Participants were exposed to topically applied 0.25% LDE225 cream twice daily for 6 weeks.
  Interventions: Drug: LDE225 0.25%
- LDE225 0.75% [Part II] (Active Comparator): Participants were exposed to topically applied 0.75% LDE225 cream twice daily where some basal cell carcinomas (BCCs) were teated for 6 weeks and some BCCs were treated for 9 weeks.
  Interventions: Drug: LDE225 0.75%

INTERVENTIONS:
Drug: Vehicle — Placebo cream
  Arms: Vehicle cream (applied in parallel with LDE225 [Part I]
Drug: LDE225 0.25%
  Arms: LDE225 0.25% [Part II]
Drug: LDE225 0.75%
  Arms: LDE225 (applied in parallel with vehicle) [Part I]; LDE225 0.75% [Part II]

SUMMARY:
Part I was a double-blind, randomized, vehicle-controlled Proof of Concept (PoC) study to evaluate the safety, local tolerability, pharmacokinetics and pharmacodynamics of multiple topical administrations of LDE225 (a specific Smoothened inhibitor) on skin basal cell carcinomas in Gorlin's syndrome patients.

Following a 21-day screening period, patients were exposed to multiple doses of topically applied LDE225 twice daily for 4 weeks in a double-blind manner. The patients returned weekly for visits where each BCC was clinically evaluated and digital photographs taken. Local safety and tolerability was also assessed. After the last application of treatment, biopsies were taken from treated (both vehicle and LDE225) BCCs (three per patient) for histology, biomarker evaluation and for pharmacokinetics (skin exposure). In addition, a biopsy from LDE225-treated uninvolved perilesional skin was taken for pharmacokinetic evaluation. In total, 4 biopsies were taken: 2 for histology and biomarker and 2 for PK.

Part II of this study consisted of a 21-day screening period, a baseline period (directly before commencing the treatment period) and a treatment period of 6 or 9 weeks, depending on randomization. A clinical assessment was performed on site on the last treatment day and if a full clinical response had been observed, approximately 3 weeks after the last treatment an excision of the BCC(s) would have been performed. The study completion visit occurred either 1 week after the excision (when this visit was planned) or 1 week after the last treatment. For a subset of patients, skin biopsies were collected on the last treatment day and an excision of a BCC was also performed at that same visit.

ELIGIBILITY:
Inclusion Criteria:

- Patients with multiple basal cell carcinomas and Gorlin syndrome, or patients with multiple basal cell carcinomas and a mutation in the PTCH1 gene at chromosome 9q22.3

Exclusion Criteria:

* Previous treatment of the BCC's that are selected for treatment.
* Any systemic treatment which is known to affect BCCs esp. cytostatic treatments, retinoids and photodynamic treatments.

Other protocol defined Incl./Excl. criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-07; Primary Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Austria (2):
  - Novartis Investigative Site, Graz
  - Novartis Investigator Site, Vienna
- Novartis Investigative Site, Zurich, Switzerland

RESULTS

PARTICIPANT FLOW:
Groups:
- All Part I Participants: Participants were exposed to both topically applied 0.75% LDE225 cream and LDE225 vehicle cream twice daily for 28 days where each treatment was randomized to two different test areas on each participant.
  LDE225 0.75%
- LDE225 0.25% [Part II]: Participants were exposed to topically applied 0.25% LDE225 cream twice daily for 6 weeks.
  LDE225 0.25%
- LDE225 0.75% [Part II]: Participants were exposed to topically applied 0.75% LDE225 cream twice daily where some basal cell carcinomas (BCCs) were treated for 6 weeks and some BCCs were treated for 9 weeks.
  LDE225 0.75%
Period: Overall Study
Arm/Group | All Part I Participants | LDE225 0.25% [Part II] | LDE225 0.75% [Part II]
Started | 8 | 3 | 7
Completed | 8 | 3 | 6
Not Completed | 0 | 0 | 1
Not completed — Abnormal laboratory value | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | All Part I Participants | LDE225 0.25% [Part II] | LDE225 0.75% [Part II] | Total
Number analyzed (Participants) | 8 | 3 | 7 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50 (13.5) | 52 (11.7) | 48 (13.4) | 50 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 3 | 8
  Male | 4 | 2 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percentage of BCCs With Complete and at Least Partial Clinical Clearance
Description: Clinical response parameters were defined as (i) complete response (i.e., there is no longer any visible evidence of a lesion consistent with BCC at this site), (ii) partial response (i.e., although a BCC still remains at this site, it has demonstrated a visible decrease in size compared with baseline), and (iii) no response / worsening (i.e., the BCC has not demonstrated any visible decrease in size compared with baseline).
Time Frame: 4 weeks, 6 weeks, 9 weeks
Population: All participants were analyzed.
Measure: Number; unit: Percentage of BCCs
Units Other Than Participants: Tumors (BCCs)
Groups:
- LDE225 (Applied in Parallel With Vehicle) [Part I]: Participants were exposed to both topically applied 0.75% LDE225 cream and LDE225 vehicle cream twice daily for 28 days where each treatment was randomized to two different test areas on each participant.
  LDE225 0.75%
Arm/Group | LDE225 (Applied in Parallel With Vehicle) [Part I] | Vehicle Cream (Applied in Parallel With LDE225 [Part I] | LDE225 0.25% [Part II] | LDE225 0.75% [Part II]
Number analyzed (Participants) | 8 | 8 | 3 | 7
Number analyzed (Tumors (BCCs)) | 13 | 14 | 12 | 22
Percentage of BCCs
  Week 4, at least partial | 92 | 7 | 83 | 77
  Week 4, complete | 23 | 0 | 0 | 0
  Week 6, at least partial | NA — Treatment duration for Part I was 4 weeks only. | NA — Treatment duration for Part I was 4 weeks only. | 83 | 96
  Week 6, complete | NA — Treatment duration for Part I was 4 weeks only. | NA — Treatment duration for Part I was 4 weeks only. | 0 | 0
  Week 9, at least partial (LDE 0.75%, n=10) | NA — Treatment duration for Part I was 4 weeks only. | NA — Treatment duration for Part I was 4 weeks only. | NA — Treatment duration for Part II at LDE225 0.25% was 6 weeks only. | 100
  Week 9, complete (LDE 0.75%, n=10) | NA — Treatment duration for Part I was 4 weeks only. | NA — Treatment duration for Part I was 4 weeks only. | NA — Treatment duration for Part II at LDE225 0.25% was 6 weeks only. | 0

2. Secondary Outcome: Change From Baseline in Tumor Measurements (Part I)
Description: Measurement of the tumor size, volume and color by standardized digital photography, using dermatoscopic, macroscopic and 3D images of the BCCs was done by participant where if a participant had more than one tumor, for each of these tumors, the change from baseline was calculated (% change). From these values, the mean was calculated to get only one result per participant. Then for all the participants (n=8 both for LDE and vehicle), the mean was calculated. Photographic analysis was conducted by QuantifiCare. The volume of a lesion was measured with a special device, the "3D LIFEVIZ Micro system", which uses a lens splitter to produce two images of the skin surface, captured at the same time, with viewing angle differences close to human vision. A stereovision algorithm is then applied to reconstruct and quantitatively analyze the skin surface in 3D. A negative change from baseline indicates improvement.
Time Frame: 4 weeks
Population: All part I participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: Percent change in tumor measurement
Arm/Group | LDE225 (Applied in Parallel With Vehicle) [Part I] | Vehicle Cream (Applied in Parallel With LDE225 [Part I]
Number analyzed (Participants) | 8 | 8
Percent change in tumor measurement
  2D surface area | -38.4 (24.82) | 9.6 (6.75)
  3D surface area | -35.3 (19.68) | 7.0 (16.86)
  Height | -32.3 (25.51) | -13.2 (12.47)
  Redness | -4.8 (16.47) | 1.2 (6.99)
  Total volume | -53.4 (30.85) | -9.9 (17.21)

3. Secondary Outcome: Change From Baseline in Tumor Measurements (Part II)
Description: Measurement of the tumor size, volume and color by standardized digital photography, using dermatoscopic, macroscopic and 3D images of the BCCs was done by participant where if a participant had more than one tumor, for each of these tumors, the change from baseline was calculated (% change). From these values, the mean was calculated to get only one result per participant. Then for all the participants (n=8 both for LDE and vehicle), the mean was calculated.. Photographic analysis was conducted by QuantifiCare. The volume of a lesion was measured with a special device, the "3D LIFEVIZ Micro system", which uses a lens splitter to produce two images of the skin surface, captured at the same time, with viewing angle differences close to human vision. A stereovision algorithm is then applied to reconstruct and quantitatively analyze the skin surface in 3D. A negative change from baseline indicates improvement.
Time Frame: 4 weeks, 6 weeks, 9 weeks
Population: Part II participants with evaluable data (n=3,6) were included in the analysis.
Measure: Mean (Standard Deviation); unit: percent change in tumor measurement
Groups:
- LDE225 0.75% [Part II]: Participants were exposed to topically applied 0.75% LDE225 cream twice daily where some basal cell carcinomas (BCCs) were treated for 6 weeks and some BCCs were treated for 9 weeks.
Arm/Group | LDE225 0.25% [Part II] | LDE225 0.75% [Part II]
Number analyzed (Participants) | 3 | 6
percent change in tumor measurement
  2D surface, week 4 | -10.7 (16.81) | -22.2 (40.43)
  2D surface, week 6 | -36.3 (12.51) | -28.5 (43.64)
  2D surface area, week 9 | NA (NA) — Treatment duration for the LDE225 0.25% arm was 6 weeks only. | -26.0 (41.57)
  3D surface area , week 4 | -19.3 (4.62) | -26.9 (33.29)
  3D surface area, week 6 | -31.7 (19.03) | -35.2 (30.51)
  3D surface area, week 9 | NA (NA) — Treatment duration for the LDE225 0.25% arm was 6 weeks only. | -41.5 (30.05)
  Total volume, week 4 | -19.3 (27.82) | -43.4 (36.25)
  Total volume, week 6 | -35.2 (37.99) | -60.7 (22.11)
  Total volume, week 9 | NA (NA) — Treatment duration for the LDE225 0.25% arm was 6 weeks only. | -61.3 (31.18)

4. Secondary Outcome: Change From Baseline in Tumor Measurements (by Tumor) (Part I)
Description: Measurement of the tumor size, volume and color by standardized digital photography, using dermatoscopic, macroscopic and 3D images of the BCCs. Photographic analysis was conducted by QuantifiCare. The volume of a lesion was measured with a special device, the "3D LIFEVIZ Micro system", which uses a lens splitter to produce two images of the skin surface, captured at the same time, with viewing angle differences close to human vision. A stereovision algorithm is then applied to reconstruct and quantitatively analyze the skin surface in 3D. A negative change from baseline indicates improvement.
Time Frame: 4 weeks
Population: All part I participants were included in this analysis.
Measure: Mean (Standard Deviation); unit: Percent change in tumor measurement
Units Other Than Participants: tumors (BCCs)
Arm/Group | LDE225 (Applied in Parallel With Vehicle) [Part I] | Vehicle Cream (Applied in Parallel With LDE225 [Part I]
Number analyzed (Participants) | 8 | 8
Number analyzed (tumors (BCCs)) | 13 | 14
Percent change in tumor measurement
  2D surface area | -40.8 (24.85) | 10.6 (10.52)
  3D surface area | -34.5 (21.36) | 8.7 (20.41)
  Height | -32.0 (26.97) | -12.7 (18.93)
  Redness | -2.0 (22.50) | 1.2 (7.42)
  Total volume | -49.8 (33.68) | -9.1 (35.24)

5. Secondary Outcome: Change From Baseline in Tumor Measurements (by Tumor) (Part II)
Description: as for outcome 4
Time Frame: 4 weeks, 6 weeks, 9 weeks
Population: Part II participants with evaluable data (n=3,6) were included in the analysis.
Measure: Mean (Standard Deviation); unit: Percent change in tumor measurement
Units Other Than Participants: Tumors (BCCs)
Arm/Group | LDE225 0.25% [Part II] | LDE225 0.75% [Part II]
Number analyzed (Participants) | 3 | 6
Number analyzed (Tumors (BCCs)) | 12 | 22
Percent change in tumor measurement
  2D surface area, week 4 | -10.7 (24.23) | -24.1 (30.69)
  2D surface area, week 6 (LDE 0.75%, n=21) | -36.3 (21.52) | -33.3 (32.42)
  2D surface area, week 9 (LDE 0.75%, n=10) | NA (NA) — Treatment duration for the LDE225 0.25% arm was 6 weeks only. | -25.5 (35.71)
  3D surface area, week 4 | -19.3 (30.58) | -23.1 (28.41)
  3D surface area, week 6 (LDE 0.75%, n=21) | -31.7 (31.19) | -33.2 (23.63)
  3D surface area, week 9 (LDE 0.75%, n=10) | NA (NA) — Treatment duration for the LDE225 0.25% arm was 6 weeks only. | -38.0 (27.97)
  Total volume, week 4 | -19.3 (57.85) | -38.3 (39.75)
  Total volume, week 6 (LDE 0.75%, n=21) | -35.2 (60.52) | -56.8 (23.70)
  Total volume, week 9 (LDE 0.75%, n=10) | NA (NA) — Treatment duration for the LDE225 0.25% arm was 6 weeks only. | -58.0 (37.24)

6. Primary Outcome: Number of Participants With at Least Partial Clinical Clearance (Part I)
Description: as for outcome 1
Time Frame: day 8, day 15, day 22, day 29
Population: All part I participants were included in the analysis.
Measure: Number; unit: Number of participants
Arm/Group | LDE225 (Applied in Parallel With Vehicle) [Part I] | Vehicle Cream (Applied in Parallel With LDE225 [Part I]
Number analyzed (Participants) | 8 | 8
Number of participants
  Day 8 | 5 | 1
  Day 15 | 7 | 2
  Day 22 | 8 | 1
  Day 29 | 8 | 1

ADVERSE EVENTS:
Groups:
- All Part I Participants: Participants were exposed to both topically applied 0.75% LDE225 cream and LDE225 vehicle cream twice daily for 28 days where each treatment was randomized to two different test areas on each participant.
- 0.25% LDE225 [Part II]: Participants were exposed to topically applied 0.25% LDE225 cream twice daily for 6 weeks.
- 0.75% LDE225 [Part II]: Participants were exposed to topically applied 0.75% LDE225 cream twice daily where some basal cell carcinomas (BCCs) were treated for 6 weeks and some BCCs were treated for 9 weeks.
Arm/Group | All Part I Participants | 0.25% LDE225 [Part II] | 0.75% LDE225 [Part II]
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/3 | 1/7
Other Adverse Events (participants affected / at risk) | 7/8 | 2/3 | 5/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Part I Participants (N=8) | 0.25% LDE225 [Part II] (N=3) | 0.75% LDE225 [Part II] (N=7)
HEPATIC ENZYME INCREASED (Investigations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Part I Participants (N=8) | 0.25% LDE225 [Part II] (N=3) | 0.75% LDE225 [Part II] (N=7)
EXTERNAL EAR INFLAMMATION (Ear and labyrinth disorders) | 0 | 0 | 1
CONJUNCTIVITIS (Eye disorders) | 0 | 0 | 1
FATIGUE (General disorders) | 0 | 0 | 1
INFECTION (Infections and infestations) | 0 | 0 | 1
NASOPHARYNGITIS (Infections and infestations) | 1 | 0 | 0
ARTHROPOD STING (Injury, poisoning and procedural complications) | 1 | 0 | 0
INJURY CORNEAL (Injury, poisoning and procedural complications) | 0 | 0 | 1
LIMB INJURY (Injury, poisoning and procedural complications) | 1 | 0 | 0
BLOOD CHOLESTEROL INCREASED (Investigations) | 1 | 0 | 0
BLOOD GLUCOSE INCREASED (Investigations) | 1 | 0 | 0
BLOOD TRIGLYCERIDES INCREASED (Investigations) | 1 | 0 | 0
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0
GLUCOSE URINE PRESENT (Investigations) | 1 | 0 | 0
HAEMATOCRIT DECREASED (Investigations) | 0 | 1 | 0
HAEMOGLOBIN DECREASED (Investigations) | 0 | 1 | 0
WHITE BLOOD CELLS URINE POSITIVE (Investigations) | 2 | 0 | 0
IRON DEFICIENCY (Metabolism and nutrition disorders) | 0 | 1 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
SKIN FISSURES (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 4 | 0 | 1
URTICARIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.